CLINICAL TRIAL: NCT05630092
Title: Comparison of the Standard 6-Minute Maximal Speed Walk Test Against a 6-Minute Normal Speed Walk Test as an Alternative and More Accurate Assessment for Ambulatory Oxygen Requirement.
Brief Title: Comparing 6-Minute Walk Tests for Ambulatory Oxygen Assessment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hampshire Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2022 SPON-HG-0922; 306758 (Registry Identifier: IRAS Project ID)
Record Dates: First submitted 2022-09-09; First posted 2022-11-29 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-02

CONDITIONS: Respiratory Disease
MeSH Terms: conditions — Respiration Disorders | interventions — Walk Test

STUDY DESIGN:
Intervention Model Description: Perform test A followed by test B (randomised order)
Who Masked: Care Provider
Masking Description: Results from the modified walk test will not be provided to the medical team prescribing ambulatory oxygen assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maximal then Normal Speed Walk Test (Active Comparator): Maximal speed walking test (Max_6MWT) followed by normal speed walking test (Nor_6MWT).
  Interventions: Diagnostic Test: Maximal 6-minute Walk Test (Max_6MWT); Diagnostic Test: Normal speed 6-minute Walk Test (Nor_6MWT)
- Normal then Maximal Speed Walk Test (Active Comparator): Normal speed walking test (Nor_6MWT) followed by Maximal speed walking test (Max_6MWT)
  Interventions: Diagnostic Test: Maximal 6-minute Walk Test (Max_6MWT); Diagnostic Test: Normal speed 6-minute Walk Test (Nor_6MWT)

INTERVENTIONS:
Diagnostic Test: Maximal 6-minute Walk Test (Max_6MWT) — Instructions given to perform the walk test following the international guidelines using the phrase 'as far as you can'.
Diagnostic Test: Normal speed 6-minute Walk Test (Nor_6MWT) — Instructions given to perform the walk test following the international guidelines except using the phrase 'at a speed you would normally walk'.

SUMMARY:
Patients with lung disease who report breathlessness on exertion are often referred for a 6MWT. Due to the nature of the 6MWT (hereon referred to as a Max-6MWT), patients are required to walk as far as they can in 6 minutes. This may lead to an inaccurate assessment of their requirement for ambulatory oxygen as this form of exercise may not correspond to their normal daily activities.

In this study, patients who are routinely referred for a Max-6MWT to investigate possible exercise-induced hypoxaemia will be invited to perform an additional walking test which is performed at their normal walking speed, referred here on in as a Nor_6MWT. We hypothesise that performing a Nor_6MWT will provide a more accurate assessment of a patients' oxygen requirement, primarily from their oxygen desaturation during the test.

DETAILED DESCRIPTION:
Patients with lung disease who report breathlessness on exertion are often referred for a 6MWT. During this test patients are asked to walk up and down a corridor (or other flat area) for six minutes whilst their blood oxygen levels and heart rate are non-invasively measured using a pulse oximeter (finger probe) and the distance walked is measured. In addition, a questionnaire that obtains a Borg Score measures the patients perceived breathlessness and leg muscle fatigue both before and immediately following the test.

Due to the nature of the 6MWT (hereon referred to as a Max-6MWT), patients are required to walk as far as they can in 6 minutes. This may lead to an inaccurate assessment of their requirement for ambulatory oxygen as this form of exercise may not correspond to their normal daily activities. It may also not accurately measure the normal changes in oxygen saturation (or desaturation) that occurs in these patients during their normal daily activities (such as walking to the shops, walking up the stairs, gardening).

In this study, patients who are routinely referred for a Max-6MWT to investigate possible exercise-induced hypoxaemia will be invited to perform an additional walking test which is performed at their normal walking speed, referred here on in as a Nor_6MWT. We hypothesise that performing a Nor_6MWT will provide a more accurate assessment of a patients' oxygen requirement, primarily from their oxygen desaturation during the test.

ELIGIBILITY:
Inclusion Criteria:

* Referred for a standard 6-minute walk test
* Has the capacity to give informed consent
* Is aged between 18 and 90

Exclusion Criteria:

* Lack of capacity to provide informed consent
* Poor peripheral perfusion that prevents an accurate measurement of SpO2
* Contraindicated to perform a Max_6MWT as indicated in the standard HHFT 6MWT SO

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Average drop in SpO2 from baseline to nadir | During the walk test
  Continuous monitoring of SpO2 will allow for the measurement in the drop from baseline to the lowest point (nadir) during the test. Between the walk tests, the average drop will be calculated and compared.

SECONDARY OUTCOMES:
Is there a difference in the time taken to reach nadir in SpO2? | During the walk test
  The time from the start of the test and the lowest (nadir) SpO2 will be recorded and compared between the walk tests.
Is there a difference in the absolute nadir SpO2 between maximal and normal walking.speed? | During the walk test
  The absolute lowest (nadir) SpO2 value will be recorded during each test and compared.

OTHER OUTCOMES:
At what time does the nadir in SpO2 occur during a Nor_6MWT | During the walk test
  Measurement of the time taken to reach nadir in SpO2 will be recorded to help justify the length of the walk test

CONTACTS AND LOCATIONS:
Overall Officials: Harry Griffin, PhD, Principal Investigator — Hampshire Hospitals NHS Foundation Trust; Michael J Hughes, PhD, Principal Investigator — Hampshire Hospitals NHS Foundation Trust
Locations (1):
- Hampshire Hospitals NHS Foundation Trust, Basingstoke, United Kingdom

IPD SHARING:
Plan to Share IPD: No